CLINICAL TRIAL: NCT04332770
Title: Clinical Application of Continuous Monitoring Data for Biosignals by Commercially Available Wearable Devices in the Patients With Hypothyroidism
Brief Title: Biosignals by Wearable Devices in Hypothyroidism
Acronym: Hypo_AT
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Hoon Moon, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1906/547-304
Record Dates: First submitted 2019-12-13; First posted 2020-04-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothyroid group: Patients with differentiated thyroid carcinoma underwent total thyroidectomy Patients who are planned to withdraw their levothyroxine for radioactive iodine therapy Biosignals will be monitored continuously using Fitbit devices
  Interventions: Other: levothyroxine withdrawal
- Control group: Patients with differentiated thyroid carcinoma underwent total thyroidectomy Patients who are planned to get rhTSH (not to withdraw their levothyroxine) for radioactive iodine therapy Biosignals will be monitored continuously using Fitbit devices

INTERVENTIONS:
Other: levothyroxine withdrawal — All participants of this study are decided to get radioactive iodine therapy using levothyroxine withdrawal or human recombinant TSH injection prior to the study enrollment. That decision is independent with this study protocol. This study just collect continuous bio signals using wearable devices in the patients undergoing two different preparation methods for radioactive iodine therapy. That is why this study is an observational cohort study.
  Groups: Hypothyroid group

SUMMARY:
This is a prospective observational cohort study. Monitoring continuous biosignals using wearable devices in thyroid cancer patients who are planned to withdraw their levothyroxine for radioactive iodine therapy. Through this, bio signals can be collected in the subjects in hypothyroid status. Physical activity, heart rate, and sleep data will be collected during the study period.

DETAILED DESCRIPTION:
A prospective observational cohort study including two groups.

Hypothyroid group:

Patients with differentiated thyroid carcinoma underwent total thyroidectomy Patients who are planned to withdraw their levothyroxine for radioactive iodine therapy Biosignals will be monitored continuously using Fitbit devices

Control group:

Patients with differentiated thyroid carcinoma underwent total thyroidectomy Patients who are planned to get rhTSH (not to withdraw their levothyroxine) for radioactive iodine therapy Biosignals will be monitored continuously using Fitbit devices Thyroid hormone levels and continuously collected bio signals including activity, heart rate, and sleep data will be obtained during study period.

Association between thyroid status and bio signals will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with differentiated thyroid carcinoma underwent total thyroidectomy
* Patients who are planned to get radioactive iodine therapy
* Patients who are able to use wearable device and smartphones

Exclusion Criteria:

* Patients who are not able to use wearable device and smartphones
* Patients who are maintaining drugs affecting heart rate
* Patients who have any other disease which can affect biosignals

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with differentiated thyroid carcinoma underwent total thyroidectomy Patients who are planned to get radioactive iodine therapy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
physical activity (steps) | throughout the study period average 4 months
  steps data measured by wearable device, collected and recorded in 1 min increment
heart rate (beats) | throughout the study period average 4 months
  heart rate data measured by wearable device, collected and recorded in 1 min increment
free T4 level (ng/dL) | baseline (visit 1)
  thyroid hormone level
free T4 level (ng/dL) | after 2 to 3 months (visit 2)
  thyroid hormone level
free T4 level (ng/dL) | after 3 to 4 months (visit 3)
  thyroid hormone level
Zulewski hypothyroidism score ( point) | baseline (visit 1)
  Scoring system to evaluate hypothyroid symptoms and signs
Zulewski hypothyroidism score ( point) | after 2 to 3 months (visit 2),
  Scoring system to evaluate hypothyroid symptoms and signs
Zulewski hypothyroidism score ( point) | after 3 to 4 months (visit 3)
  Scoring system to evaluate hypothyroid symptoms and signs
TSH level (mIU/L) | baseline (visit 1)
  thyroid stimulating hormone level
TSH level (mIU/L) | after 2 to 3 months (visit 2)
  thyroid stimulating hormone level
TSH level (mIU/L) | after 3 to 4 months (visit 3)
  thyroid stimulating hormone level

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hoon Moon, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No